CLINICAL TRIAL: NCT03096639
Title: Percutaneous Temporary Placement of a Phrenic Nerve Stimulator for Diaphragm Pacing
Acronym: RESCUE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lungpacer Medical Inc. (Industry)
Collaborators: Syntactx (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-200
Record Dates: First submitted 2017-03-15; First posted 2017-03-30 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Ventilator Induced Diaphragm Dysfunction
Keywords: Diaphragm atrophy; VIDD; Weaning failure

STUDY DESIGN:
Intervention Model Description: 1:1 randomization of treatment and control group
Who Masked: Outcomes Assessor
Masking Description: The ultrasound core lab reviewers will be blinded to study allocation groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Diaphragm Pacing Therapy DPTS (Active Comparator): Diaphragm Pacing intervention will be conducted 2x a day using the Diaphragmatic Pacing Therapy System (DPTS). The DPTS includes the Lungpacer IntraVenous Electrode Catheter (LIVE Catheter) which is inserted temporarily into the left subclavian vein, the Lungpacer Control Unit (LCU external unit) and an intermediate cable that connects the LCU to the LIVE Catheter.
  Interventions: Device: Diaphragmatic Pacing Therapy DPTS
- Control Group (No Intervention): Standard of care treatment of weaning failure, no intervention is involved in this control group.

INTERVENTIONS:
Device: Diaphragmatic Pacing Therapy DPTS — Subjects will undergo DPTS 2 times a day until successfully extubated with no reintubation within 48 hours.
  Other Names: DPTS; LIVE Catheter
  Arms: Diaphragm Pacing Therapy DPTS

SUMMARY:
A randomized clinical trial to investigate the use of the temporary Diaphragm Pacing Therapy System (DPTS) to rehabilitate the diaphragm in mechanically ventilated patients who have failed at least two weaning attempts. The goal is to strengthen and rehabilitate the diaphragm to liberate the patient more quickly from mechanical ventilation.

DETAILED DESCRIPTION:
Mechanical ventilation (MV) is a life saving technology but can also cause damage to the lungs and diaphragm such as ventricular induced diaphragmatic dysfunction (VIDD). Research has shown that after being on mandatory MV and sedated the diaphragm begins to atrophy within as short as 18 hours. The Lungpacer Diaphragm Pacing Therapy System (DPTS) is a temporary therapy that consists of the Lungpacer IntraVenous Electrode Catheter (LIVE Catheter) and the Lungpacer Control Unit system. The LIVE Catheter is a proprietary central venous catheter that incorporates pacing electrodes in strategic areas that align with the left and right phrenic nerves. The LIVE Catheter can also be used for fluid delivery like any other central venous catheter. The randomized clinical trial will investigate the safety, effectiveness and performance of the Lungpacer DPTS. By stimulating the diaphragm through daily therapy sessions, with the intention of exercising and rehabilitating the diaphragm muscle so the patient may be able to be more quickly liberated from MV. The patient population includes those who have been mechanically ventilated for greater than or equal to 96 hours (4days), have failed two or more spontaneous breathing trials (SBT), and were not hypervolemic during the latest spontaneous breathing trial. Patients must have resolution of the initial indication for placement on mechanical ventilation before entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* have been mechanically ventilated for > or = to 96 hours (4 days), and
* have satisfied the Readiness-to-Wean criteria and
* have failed at least two VLTs, one of which is the study specific VLT.

Exclusion Criteria:

* currently on extracorporeal membrane oxygenation (ECMO);
* weaning failure due to hypervolemia;
* medical history or known anatomy that prevents insertion of the LIVE Catheter into the left subclavian vein;
* currently being treated with neuromuscular blockade;
* clinically overt congestive heart failure that is preventing weaning;
* pre-existing neuromuscular diseases that could affect the respiratory muscles;
* pre-existing severe chronic pulmonary fibrosis;
* pleural effusions occupying greater than one third of the pleural space on either side;
* BMI > or = 40;
* known or suspected phrenic nerve paralysis;
* any electrical device (implanted or external) that may be prone to interaction with or interference from the Lungpacer DPTS including neurological pacing/stimulator devices, cardiac pacemakers and defibrillators;
* prior bacteremia reported within the last 48 hours;
* current hemodynamic instability, sepsis or septic shock;
* terminally ill with 6 months or less life expectancy or not committed to full care;
* known or suspected to be pregnant or lactating; and
* currently being treated in another clinical trial studying an experimental treatment that could affect the study primary outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-12-29 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Proportion successfully weaned by 30 days for subjects randomized to Treatment (Lungpacer DPTS) as compared to subjects randomized to Control. | Patients will be allowed to stay in the study for up to 30 (+2 days of follow up for adverse events) days if not removed from mechanical ventilation sooner
  "Successfully weaned" is defined as passing the protocol-specific Ventilator Liberation Trial (VLT), or removed from MV, and not reintubated (subjects with an oral or nasal, endotracheal tube) or returned to MV (subjects with a tracheostomy) within 48 hours

SECONDARY OUTCOMES:
Days on mechanical ventilation | from randomization to 30 days
  Days on mechanical ventilation from randomization to removal from MV associated with successful weaning or Day 30, whichever comes first
Changes in diaphragmatic thickening fraction on diaphragm ultrasound | to successful weaning or on day 30 which ever comes first.
  Evaluate difference in changes in diaphragmatic thickening fraction between study allocation groups from randomization to successful weaning or on day 30 whichever comes first;
Changes in MIP | to successful weaning, or on day 30, whichever comes first.
  Change in MIP from randomization to last available measure; Change in MIP over time from randomization (baseline).
Change in MIP | to successful weaning, or on day 30 whichever comes first.
  Rate of MIP change per day from randomization (baseline) to last available measure;
Changes in RSBI | to successful weaning, or on day 30, whichever comes first
  Change in RSBI from randomization (baseline) to last available measure; Change in RSBI over time from randomization (baseline);
Change in RSBI | to successful weaning, or on day 30, whichever comes first
  Rate of RSBI change per day from randomization (baseline) to last available measure;
Mortality | on day 30
  30-day mortality

OTHER OUTCOMES:
Weaning from and re-installation of Mechanical Ventilation in both groups | from randomization to 30 days
  Cessations and re-instatements of mechanical ventilation to Day 30 or Study Exit
Tracheostomy | from randomization to 30 days
  Proportion of subjects tracheotomized from randomization to study exit
Ventilator settings | from randomization to 30 days
  Pressure Support daily, to last available measure
Ventilator settings | from randomization to 30 days
  PEEP daily, to last available measure
Ventilator settings | from randomization to 30 days
  Ventilation Mode daily, to last available measure
Ventilator settings | from randomization to 30 days
  Tidal Volume daily, to last available measure
Number of ICU admissions and discharges through D30 for both groups | from randomization to 30 days
  ICU admissions and discharges to day 30
Number of hospital admissions and discharges through D30 for both groups | from randomization to 30 days
  Hospital admissions and discharges to day 30.

CONTACTS AND LOCATIONS:
Overall Officials: Linda H Clark, BSN, Study Director — Vice President of Clinical Affairs, Lungpacer Medical, Inc.
Locations (21):
- France (7):
  - CHU Angers, Reanimation Medicale, Angers
  - Hopital Louis-Mourier, Colombes
  - CHU Montpellier, Montpellier
  - Centre Hospitalier Universitaire de Nice (CHU Nice), Nice
  - Hopital Europeen Georges-Pompidou, Paris
  - Pitie Salpetriere Hospital, Paris
  - Centre Hospitalier Universitaire CHU, Strasbourg
- Germany (14):
  - Uniklinik RWTH Aachen, Aachen
  - Heart and Diabetes Center Bad Oeynhausen, Bad Oeynhausen
  - Charite Universitatsmedizin Berlin - Mitte campus, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Universitatsklinik Dresden, Dresden
  - Universitatsmedizin Gottingen, Georg-August-Universitat, Göttingen
  - Asklepios Kliniken Hamburg GmbH - Asklepios Klinikum Harburg, Hamburg
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Med Uni-Heidelberg, Heidelberg
  - Universitätsklinikum Jena, Jena
  - Klinikum Nuernberg, Nuremberg
  - Universitatsklinikum Regensburg, Regensburg
  - Fachkrankenhaus Kloster Grafschaft, Schmallenberg
  - Wissenschaftliches Institut Bethanien fur Pneumologie e.V., Solingen

IPD SHARING:
Plan to Share IPD: Undecided
Only investigators participating in this clinical trial will be able to see final de-identified participant data at the completion of the study and it will be available through the clinical research organization (CRO).

REFERENCES:
- [Background] Evans D, Shure D, Clark L, Criner GJ, Dres M, de Abreu MG, Laghi F, McDonagh D, Petrof B, Nelson T, Similowski T. Temporary transvenous diaphragm pacing vs. standard of care for weaning from mechanical ventilation: study protocol for a randomized trial. Trials. 2019 Jan 17;20(1):60. doi: 10.1186/s13063-018-3171-9. PMID 30654837
- [Result] Dres M, de Abreu MG, Merdji H, Muller-Redetzky H, Dellweg D, Randerath WJ, Mortaza S, Jung B, Bruells C, Moerer O, Scharffenberg M, Jaber S, Besset S, Bitter T, Geise A, Heine A, Malfertheiner MV, Kortgen A, Benzaquen J, Nelson T, Uhrig A, Moenig O, Meziani F, Demoule A, Similowski T; RESCUE-2 Study Group Investigators. Randomized Clinical Study of Temporary Transvenous Phrenic Nerve Stimulation in Difficult-to-Wean Patients. Am J Respir Crit Care Med. 2022 May 15;205(10):1169-1178. doi: 10.1164/rccm.202107-1709OC. PMID 35108175